CLINICAL TRIAL: NCT05836623
Title: A Phase I Study to Assess Biodistribution of 89Zr-CB307 in PSMA+ and PSMA- Tumour Lesions (A Sub-study of CBT307-1 Study - EUDRACT 2019-004584-46)
Brief Title: A Phase I Study to Assess PSMA+ and PSMA- Tumour Lesions
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Crescendo Biologics Ltd. (Industry)
Collaborators: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CBT307-1-RL; 2021-006256-13 (EudraCT Number)
Record Dates: First submitted 2023-03-07; First posted 2023-05-01 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Advanced and/or Metastatic Solid Tumours
Keywords: Phase 1 Study; Solid Tumours; Castration-resistant prostate cancer (CRPC); Prostate Specific Membrane Antigen (PSMA); Crescendo Biologics; CD137; CB307; Humabody®; Radiolabelled CB307; 89-Zirconium; Biodistribution; HSA

STUDY DESIGN:
Intervention Model Description: Following administration of 89Zr-CB307, enrolled patients will undergo a number of PET scans where uptake of the radiolabelled drug will be assessed
Masking Description: Open-label single center non-randomised study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part A - Optimisation Phase (Experimental): Following administration of 89Zr-CB307, patients will undergo PET scans The timing of the scans and CB307 dose administration will be determined by the Optimisation Review Committee (ORC)
  Interventions: Drug: Radiolabelled CB307; Drug: CB307
- Part B - Expansion phase (Experimental): 89Zr-CB307 PET scanning will be performed based on the optimal dosing and timing determined in Part A by the Optimisation Review Committee (ORC)
  Interventions: Drug: Radiolabelled CB307; Drug: CB307

INTERVENTIONS:
Drug: Radiolabelled CB307 — CB307 radiolabelled with 89-Zirconium (89Zr CB307): drug product is formulated at a concentration of 1 mg/mL (37 MBq)
  Other Names: 89Zr-CB307
Drug: CB307 — Trispecific Humabody® targeting CD137, prostate specific membrane antigen and human serum albumin

SUMMARY:
CB307 is a trispecific Humabody® targeting CD137; PSMA; and human serum albumin (HSA) undergoing Phase 1 assessment in patients with PSMA+ solid tumours. This sub study will assess the biodistribution of radiolabelled CB307 in patients with advanced and/or metastatic solid tumours that are PSMA+.

DETAILED DESCRIPTION:
Phase 1, Open-label, single centre, non-randomised study during which, enrolled patients will undergo a number of PET scans following administration of 89Zr-CB307, in order to assess the uptake of the radiolabelled drug. A post-treatment tumour biopsy for the assessment of PSMA expression will also be taken, if medically feasible, after the last PET scan.

The sub-study consists of 2 parts: an Optimisation Phase (Part A) and an Expansion Phase (Part B).

In Part A, both 89Zr-CB307 and CB307 will be administered to patients. The timing of the scans, post-dose tumour biopsy and CB307 dose will be optimised as determined by the Optimisation Review Committee (ORC).

In Part B (Expansion Phase), 89Zr-CB307 PET scanning will be performed based on the optimal dosing and timing determined in Part A.

The sub-study will continue for 7 days after the tracer injection. Patients will then be enrolled into the main study and will receive Cycle 1 Day 1 (C1D1) CB307 treatment according to the main study protocol.

ELIGIBILITY:
Inclusion Criteria:

* Capable of understanding the written informed consent.
* Aged at least 18 years.
* Not amenable to standard of care.
* ECOG PS of 0 or 1.
* Documented histologically confirmed diagnosis of PSMA+ advanced or metastatic solid tumours.
* Has radiologically measurable disease per RECIST v1.1 or elevated serum PSA for castration resistant prostate cancer patients with only bone metastases.
* Adequate organ function.
* Willing to have a biopsy sample taken immediately after the last PET scan before initiation of the main study.

Exclusion Criteria:

* Subjects with autoimmune disease or regular immunosuppressants.
* Has discontinued from anti-CTLA 4, anti-PD1 or anti-PD-L1 antibody because of intolerable toxicity.
* Has brain metastasis including leptomeningeal metastasis or primary brain tumour.
* Has current or history of CNS disease.
* Has known active infection.
* Biopsy cannot be safely obtained after the last PET scan, and not provided their consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2022-12-20 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Assessment of the safety of 89Zr-CB307 by assessing incidence of adverse events following administration of 89Zr-CB307. | Throughout study completion, up to 8 months from first patient recruited.
  Incidence (frequency and severity) of adverse events following administration of 89Zr-CB307 assessed by CTCAE version 5.0
Assessment of 89Zr-CB307 uptake by PET scan by measuring maximum standardized uptake value in the tumour lesions. | Throughout study completion, up to 8 months from first patient recruited.
  SUVpeak - maximum standardized uptake value.
Assessment of 89Zr-CB307 uptake by PET scan by measuring mean standardized uptake value in the tumour lesions. | Throughout study completion, up to 8 months from first patient recruited.
  SUVmean - mean standardized uptake value.
Assessment of 89Zr-CB307 uptake by PET scan by measuring percentage of injected dose per gram of tissue in the tumour lesions. | Throughout study completion, up to 8 months from first patient recruited.
  %ID/g - percentage of injected dose per gram.

CONTACTS AND LOCATIONS:
Overall Officials: Julia Tilson, Study Director — Crescendo Biologics Limited
Locations (1):
- University Medical Center Groningen,, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No